CLINICAL TRIAL: NCT05777967
Title: A Phase 3 Single-arm Multicenter Study of FF-31501 in Meniscus Tear Patients
Brief Title: Efficacy and Safety of FF-31501 in Meniscus Tear Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF31501JP301
Record Dates: First submitted 2023-02-08; First posted 2023-03-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Meniscus Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Biological: human autologous synovial stem cells

INTERVENTIONS:
Biological: human autologous synovial stem cells — A single injection of 1.5 to 9.0 x 10^7 human autologous synovial stem cells under arthroscopy

SUMMARY:
A single-arm, multi-center study to verify that knee joint function at 52 weeks after injection of FF-31501 is better than at screening in patients with meniscus tear who are eligible for meniscectomy .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected meniscal flap tear
2. Patients with knee pain
3. Patients with one or more of the following symptoms

   * Feeling stuck in the knee・Instability of the knee
   * Knee range of motion impairment
   * Knee joint edema
4. Other

Exclusion Criteria:

1. Patients with poor knee alignment
2. Patients who underwent meniscus surgery or platelet rich plasma therapy
3. Patients with or history of knee ligament injury
4. Diabetic patients with poor glycemic control
5. Patients with the following complications and poor general condition

   * Severe cardiovascular disease
   * Severe liver disease
   * Severe renal dysfunction
   * Severe anemia・uncontrolled mental illness
   * Other diseases for which sudden change or worsening of symptoms can be expected during study participation
6. Patients who are pregnant or possibly pregnant and/or breast-feeding, or patients planning to become pregnant during the study period
7. Other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Lysholm score | Screening up to 52 weeks
  It consists of items that measure: pain, instability, locking, swelling, limp, stair climbing, squatting, and need for support. Lowest and highest scores are 0 and 100 (better), respectively.

SECONDARY OUTCOMES:
Arthroscopic assessment of the meniscus | Meniscus repair up to 52 weeks
  The structure and function of the repaired meniscus will be assessed in terms of the presence, stability, and smoothness of the meniscus by arthroscopic imaging and MRI.
Knee injury and osteoarthritis outcome score (KOOS) | Screening up to the Day before injection,4,12,24 and 52 weeks
  The KOOS consists of five subscales; Pain, other symptoms, function in daily living (ADL), function in sport and recreation (Sport/Rec) and knee related quality of life (QOL). Lowest and highest scores are 0 and 100 (better), respectively.
Numerical Rating Scale (NRS) | Screening up to the Day before injection,4,12,24 and 52 weeks
  NRS consists of an 11-point scale to evaluate current knee pain where no pain is indicated by '0', and the worst pain imaginable by '10'.
Kellgren Lawrence | Screening up to 24 and 52 weeks
  The Kellgren and Lawrence system is a common method of classifying the severity of osteoarthritis (OA) using five grades.

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Medical corporation keimeikai Juko Osu hospital, Aichi
  - Wakamatsu Hospital of the University of OccupationalOC and Environmental Health, Fukuoka
  - Mie Prefectural General Medical Center, Mie
  - Tokyo Medical and Dental University Hospital, Tokyo